CLINICAL TRIAL: NCT05916300
Title: Diagnostic Ultrasonography in Physiotherapy as a Prevention of the Development of Complications of Post-Traumatic Ankle Conditions
Brief Title: Diagnostic Ultrasonography in Physiotherapy
Acronym: SonograPHY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Petr Routner (Other)
Responsible Party: Sponsor-Investigator, Petr Routner, Principal Investigator, Charles University, Czech Republic
Organization: Charles University, Czech Republic (Other)
Other Study IDs: 81512267
Record Dates: First submitted 2023-04-26; First posted 2023-06-23 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Ankle Sprains; Ankle Injuries; Ankle Edema; Ankle Impingement; Ankle Fractures
Keywords: Diagnostic ultrasonography; physiotherapy; post-traumatic ankle conditions; prevention
MeSH Terms: conditions — Ankle Injuries; Ankle Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard physiotherapy group: Patients will be treated with standard physiotherapy according to the recommendation of the referring physician without modification of the treatment based on the output of the diagnostic ultrasonography examination.
  Interventions: Other: Diagnostic ultrasonography-guided physiotherapy group
- Diagnostic ultrasonography-guided physiotherapy group: Patients will undergo modified treatment techniques, the application of which will be indicated based on the initial diagnostic ultrasonographic examination.
  Interventions: Other: Diagnostic ultrasonography-guided physiotherapy group

INTERVENTIONS:
Other: Diagnostic ultrasonography-guided physiotherapy group — All participants will complete free 10 outpatient 30-minute sessions. The therapy will be focused on increasing the range of motion and muscle strength, optimizing the function of the lower limbs, reducing possible complications of post-traumatic conditions in the ankle area.
  The physiotherapy procedures of the intervention group will be modified based on the initial diagnostic ultrasonography examination.

SUMMARY:
Ankle injuries are among the most common traumatological injuries of the lower limb accounting for approximately 50% of all sports injuries and 25% of musculoskeletal injuries in general. Correct initial diagnosis and proper management is important to reduce the risk of recurrent ankle instability and other complications, such as reduced range of motion, increased ligament laxity, instability, tendon enthesopathy, possible swelling, formation of calcifications, reduced load on the affected limbs while standing and walking, increased pain intensity and pain duration. To date, few studies showed that the effectiveness of physical therapy increases when it is modified based on diagnostic ultrasonography findings. Sonography is not burdensome for the patient, has high reproducibility, and enables dynamic examination and comparison of the interrelationships of individual structures.

The aim of this study is to investigate if targeted physiotherapy for post-traumatic ankle conditions designed based of diagnostic ultrasonography findings is more effective than standard physiotherapy. The study hypothesis is that in the experimental group there will be a smaller number of complications of post-traumatic ankle conditions than in the control group. If confirmed the study could have clinical implications.

DETAILED DESCRIPTION:
A randomized controlled trial

In a randomized controlled trial, patients with post-traumatic soft tissue damage in the ankle area will be randomly divided into two groups. Both groups will undergo the same number of physiotherapy sessions (10 half-hour outpatient sessions over the course of two months) and will be examined with standard clinical tests and diagnostic ultrasonography at the beginning of the program and at week 8 using a standardized protocol published by the European Society of Musculoskeletal Radiology. Both groups will undergo the same physiotherapy techniques. Their choice will be modified in the experimental group based on the current findings of diagnostic sonography, while in the control group they will be applied according to the standard procedure recommended by the physician.

Randomization

Participants meeting the entry criteria will be examined by diagnostic ultrasonography, then randomly assigned to two groups using software (https://www.randomizer.org/) and sent for an entry examination by an independent investigator. Group 1 will undergo standard physiotherapy without continuous monitoring of the course and effect of treatment with diagnostic ultrasonography. The treatment of the second group will be modified based on the current findings of the diagnostic ultrasonography. The therapeutic protocol for each patient will be given to an independent physiotherapist (the therapist will not know the details of the study) in a sealed envelope.

Study participants

Study participants will be recruited based on referrals from specialists (mainly orthopaedists or surgeons) following the entry and exclusion criteria below. When a patient meeting the criteria is detected, the specialist will offer the patient the opportunity to participate in the study, and if agreed, the patient will be sent to our workplace for an initial examination.

Sample size

A sample size of 26 patients per group (N=52) was estimated to test the difference in pain (primary outcome, scale 0-10; at 80% test power (Cohen´s d=0.8) and at the 0.05 significance level) between the intervention and control groups. We estimate that 15% of participants will not complete the study, therefore 68 patients will be enrolled in the study (34 patients in each group).

Basic statistical analysis of outcome variables

Difference in numeric variables (pain, chronic ankle instability rate, the 10 Metre Walk Test, examination of ankle dorsiflexion muscle strength) between the intervention and control groups will be tested using the two-sample t-test or Mann-Whitney Test, if normality of the data was not fulfilled. Data normality will be assessed using the Shapiro-Wilk test and visually using box and whisker plots, histograms and normal probability plots. Difference in categorical variables (the range of motion of the ankle, the presence of swelling, number of complications) will be tested using chi-square test or Fisher's exact test, if at least one expected frequency will be smaller than 5. R software will be used for analysis.

Examination

Demographic, anthropometric and anamnestic data of all participants will be recorded at the beginning of the programme (age, sex, height, weight, exercise history, injury history, including frequency of past injuries, footwear). The clinical examination will be carried out at the beginning and at the end of the therapeutic program, i.e. after two months from the start of the program.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 15 years and ≤ 65 years
* Post-traumatic conditions in the ankle area, 0 - 6 weeks after the primary injury
* Ability to undergo continuous outpatient physiotherapy treatment
* Active cooperation of the patient

Exclusion Criteria:

* Age < 15 years and > 65 years
* Serious diseases affecting effective physiotherapy (e.g. tissue damage of metabolic, degenerative, neurological or oncological origin)
* Previous ankle surgery
* Gypsum fixation

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acute post-traumatic ankle conditions
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pain level | The change from baseline to 8 weeks
  Examination using the Wong-Baker scale. The scale is used to subjectively assess pain. Pain rating scale (0-10): 0 - no pain; 2 - hurts a little; 4 - hurts a little more; 6 - hurts even more; 8 - hurts a lot; 10 - hurts the most (0 is the best value, 10 is the worst).
The range of motion of the ankle | The change from baseline to 8 weeks
  Goniometry will be performed with a stainless steel two-arm goniometer (ref. SH5103).
  Measurement of the ankle (talocrural joint) dorsiflexion range of motion: Participants will actively adduct the tip of the injured ankle while sitting on a physical therapy table. The expected range of motion with knee extension is approx. 10 degrees, with 20 degrees of knee flexion. For the evaluation, we will use a 3-point evaluation scale: 0-3 (0 - no limitation in dorsiflexion, 1 - small limitation in dorsiflexion, 2 - great limitation in dorsiflexion, 3 - no movement in dorsiflexion) (0 means the best value, 3 is the worst).
The measurement of swelling | The change from baseline to 8 weeks
  Over the course of the therapy, we will measure the swelling with a standard retractable four-inch plastic tape measure and a marking pen according to a standardized protocol. (decreasing the size of edema over time marks positive change).
Number of complications | The change from baseline to 8 weeks
  The following complications will be monitored using sonographic examination based on a standardized protocol issued by the European Society of Musculoskeletal Radiology using a 7L4BP 5-10 MHz linear probe.
  The following complications will be measured according to standardized methodologies and evaluated by comparison with the same measured parameters on the ankle of the uninjured leg: 1. greater thickness of the ligaments (anterior tibiofibular and anterior talofibular ligament); 2. the presence of exudate in the area of anterior talofibular ligament, 3. the presence of calcifications, 4. a reduction in the continuity of the ligament apparatus in the ankle or the continuity of the syndesmosis compared to the non-affected leg. A higher number means a higher number of complications.

SECONDARY OUTCOMES:
Chronic ankle instability rate | The change from baseline to 8 weeks
  The Cumberland Ankle Instability Tool (CAIT) is a simple, valid and reliable instrument for discriminating and measuring the severity of functional ankle instability. The CAIT comprises a 9-item 30-point scale questionnaire (the higher final score indicates less severe functional ankle instability). Subjects with a score of 28 or higher are unlikely to have functional ankle instability, whereas subjects with a score of 27 or lower are likely to have functional ankle instability.
Analysis of standing and walking | The change from baseline to 8 weeks
  The 10 Metre Walk Test. We will measure the gait speed, using a stopwatch and markers, a phone with a camera (the lower value means better result).
Examination of ankle dorsiflexion muscle strength | The change from baseline to 8 weeks
  The examination will be held using a microFET2 hand-held digital dynamometer (Hoggan Scientific, USA).
  The examination will be held according to a standardized protocol: Subjects will lie supine with the knee extended and ankle of the tested leg in a neutral position on the bed. Ankle dorsiflexion will be tested by placing a dynamometer over the dorsal surface of the midfoot, just proximal to the metatarsal phalangeal joints. We will measure the isometric muscle strength (in N) when the patient tries for maximum resistance against the dynamometer of the affected ankle for four seconds. A higher value of muscle strength after rehabilitation means an improvement of the condition.

CONTACTS AND LOCATIONS:
Overall Officials: Petr Routner, MSc., Principal Investigator — Department of Rehabilitation Medicine, Third Faculty of Medicine, Charles University in Prague; Kamila Řasová, PT, PhD., Study Director — Department of Rehabilitation Medicine, Third Faculty of Medicine, Charles University in Prague
Locations (1):
- Alafia-RHB, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
All data sharing terms and conditions and the nature of the relationship between the study and new user will be contained in a Data-sharing Agreement that will be issued and signed before any data are handed out. The de-identification process for each patient is to ensure anonymization of individual patient's data, in order to be able to share IPD within the terms of participant's consent and ethics committee approval.
  The study policy on sharing defines the terms of privileged use by the study team. The research team requires to be appropriately notified and acknowledged in publications and other outputs of the transferred data (or analyses conducted by the study on the new users' behalf). The Data-sharing agreement will comprehend arrangements for data destruction or secure archiving.
  It is planned that the data will be placed into an online repository (to be specified later).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The IPD will be made available from 3-months following the first publication of findings based on the data until 3 years following the first publication.
Access Criteria: The datasets will be prepared and might be reachable upon a request. The study team formally reviews access requests for proposals. The data on an exclusive basis will be made available for third party use/ the new user, which can range from direct provision of data, data analysis collaboration, and/or scientific collaboration. Also, the requester is to state the purpose for which the data are to be used.

REFERENCES:
- [Background] Fernandez WG, Yard EE, Comstock RD. Epidemiology of lower extremity injuries among U.S. high school athletes. Acad Emerg Med. 2007 Jul;14(7):641-5. doi: 10.1197/j.aem.2007.03.1354. Epub 2007 May 18. PMID 17513688
- [Background] Bergman R, Shuman VL. Acute Ankle Sprain. 2025 Aug 2. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK459212/ PMID 29083595
- [Background] Martin B. Ankle sprain complications: MRI evaluation. Clin Podiatr Med Surg. 2008 Apr;25(2):203-47, vi. doi: 10.1016/j.cpm.2007.12.004. PMID 18346591
- [Background] Faltus J, Boggess B, Bruzga R. The use of diagnostic musculoskeletal ultrasound to document soft tissue treatment mobilization of a quadriceps femoris muscle tear: a case report. Int J Sports Phys Ther. 2012 Jun;7(3):342-9. No abstract available. PMID 22666649
- [Background] Innes S, Jackson J. Musculoskeletal ultrasound imaging - An exploration of physiotherapists' interests and use in practice. Musculoskelet Sci Pract. 2019 Dec;44:102068. doi: 10.1016/j.msksp.2019.102068. Epub 2019 Sep 30. PMID 31585403
- [Background] Sconfienza LM, Adriaensen M, Albano D, Alcala-Galiano A, Allen G, Aparisi Gomez MP, Aringhieri G, Bazzocchi A, Beggs I, Chianca V, Corazza A, Dalili D, De Dea M, Del Cura JL, Di Pietto F, Drakonaki E, Facal de Castro F, Filippiadis D, Gitto S, Grainger AJ, Greenwood S, Gupta H, Isaac A, Ivanoski S, Khanna M, Klauser A, Mansour R, Martin S, Mascarenhas V, Mauri G, McCarthy C, McKean D, McNally E, Melaki K, Messina C, Miron Mombiela R, Moutinho R, Olchowy C, Orlandi D, Prada Gonzalez R, Prakash M, Posadzy M, Rutkauskas S, Snoj Z, Tagliafico AS, Talaska A, Tomas X, Vasilevska Nikodinovska V, Vucetic J, Wilson D, Zaottini F, Zappia M, Obradov M. Clinical indications for image-guided interventional procedures in the musculoskeletal system: a Delphi-based consensus paper from the European Society of Musculoskeletal Radiology (ESSR)-part VI, foot and ankle. Eur Radiol. 2022 Feb;32(2):1384-1394. doi: 10.1007/s00330-021-08125-z. Epub 2021 Aug 25. PMID 34432122
- [Background] HEROLD, I. Hodnocení bolesti a kvality analgezie u kriticky nemocných na JIP. Anesteziologie a Intenzivni Medicina. 2013; 24(6): 430-433. ISSN 12142158.
- [Background] PAZ, JC, QUINLAN, D. Acute Pain Management. Acute Care Handbook for Physical Therapists-E-Book. 2013; 7: 457-465.
- [Background] WATSON CP, BOLAND RA., REFSHAUGE KM. Measurement reliability of swelling in the acute ankle sprain. The Foot & Ankle Journal. 2008; 1(12): 4.
- [Background] Esterson PS. Measurement of ankle joint swelling using a figure of 8*. J Orthop Sports Phys Ther. 1979;1(1):51-2. doi: 10.2519/jospt.1979.1.1.51. PMID 18810189
- [Background] Hiller CE, Refshauge KM, Bundy AC, Herbert RD, Kilbreath SL. The Cumberland ankle instability tool: a report of validity and reliability testing. Arch Phys Med Rehabil. 2006 Sep;87(9):1235-41. doi: 10.1016/j.apmr.2006.05.022. PMID 16935061
- [Background] Sisto SA, Dyson-Hudson T. Dynamometry testing in spinal cord injury. J Rehabil Res Dev. 2007;44(1):123-36. doi: 10.1682/jrrd.2005.11.0172. PMID 17551866
- [Background] Yin Y, Yu Z, Wang J, Sun J. Effectiveness of the Rehabilitation Training Combined with Maitland Mobilization for the Treatment of Chronic Ankle Instability: A Randomized Controlled Trial. Int J Environ Res Public Health. 2022 Nov 20;19(22):15328. doi: 10.3390/ijerph192215328. PMID 36430049
- [Background] MCNALLY, E. Practical musculoskeletal ultrasound E-Book [online]. 2nd Edition. Churchill Livingstone, 2014. ISBN 978-1-4557-7404-3.
- [Background] SCHMITZ, Marc J.H. Musculoskeletal ultrasound of the extremity joints : technical scanning guidelines [online]. SonoSkills, 2022. ISBN 9083240304.
- [Background] BEGGS, Ian, STEFANO BIANCHI, ANGEL BUENO, MICHEL COHEN, MICHEL COURT-PAYEN, ANDREW GRAINGER, FRANZ KAINBERGER, ANDREA KLAUSER, CARLO MARTINOLI, EUGENE MCNALLY, J PHILIPO, PHILIPPE PEETRONS, MONIQUE REIJNIERSE. European Society of MusculoSkeletal Radiology Musculoskeletal Ultrasound Technical Guidelines VI. Ankle [online]. 2016 [cit. 2023-03-08]. Available at: https://essr.org/content-essr/uploads/2016/10/ankle.pdf
- [Background] Petersen EJ, Irish SM, Lyons CL, Miklaski SF, Bryan JM, Henderson NE, Masullo LN. Reliability of water volumetry and the figure of eight method on subjects with ankle joint swelling. J Orthop Sports Phys Ther. 1999 Oct;29(10):609-15. doi: 10.2519/jospt.1999.29.10.609. PMID 10560070
- [Background] Bohannon RW. Reference values for extremity muscle strength obtained by hand-held dynamometry from adults aged 20 to 79 years. Arch Phys Med Rehabil. 1997 Jan;78(1):26-32. doi: 10.1016/s0003-9993(97)90005-8. PMID 9014953
- [Background] R CORE TEAM. R Core Team 2021 R: A language and environment for statistical computing. R foundation for statistical computing. https://www.R-project.org/. R Foundation for Statistical Computing [online]. 2022, 2, 2019 [cit. 2023-01-30]. Available at: https://www.scirp.org/(S(czeh2tfqw2orz553k1w0r45))/reference/referencespapers.aspx?referenceid=3131254
- [Background] De Maeseneer M, Marcelis S, Jager T, Shahabpour M, Van Roy P, Weaver J, Jacobson JA. Sonography of the normal ankle: a target approach using skeletal reference points. AJR Am J Roentgenol. 2009 Feb;192(2):487-95. doi: 10.2214/AJR.08.1316. PMID 19155415
- [Background] Bandinelli S, Benvenuti E, Del Lungo I, Baccini M, Benvenuti F, Di Iorio A, Ferrucci L. Measuring muscular strength of the lower limbs by hand-held dynamometer: a standard protocol. Aging (Milano). 1999 Oct;11(5):287-93. doi: 10.1007/BF03339802. PMID 10631877
- See also: Goniometry: Ankle (Talocrural) Dorsiflexion - Physiopedia — https://www.physio-pedia.com/Goniometry:_Ankle_(Talocrural)_Dorsiflexion
- See also: CORE MEASURE: 10 METER WALK TEST (10mWT) — https://www.neuropt.org/docs/default-source/cpgs/core-outcome-measures/core-measure-10-meter-walk-test-(10mwt)_final.pdf
- See also: Gait Range of Motion Animation — https://www.youtube.com/watch?v=5Z6shSu96CM
- See also: microFET2 User Guide — https://www.fysiosupplies.nl/media/PDF/microFET2_BLUETOOTH_manual.pdf